CLINICAL TRIAL: NCT00139815
Title: An International, Randomized, Double-blind Study Evaluating the Efficacy and Safety of Fondaparinux Versus Enoxaparin in the Acute Treatment of Unstable Angina/Non ST-segment Elevation MI Acute Coronary Syndromes
Brief Title: Michelangelo - Oasis 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Chicago (Other); Organon (Industry); Sanofi (Industry); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103420; NCT01352169 (obsolete NCT alias)
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Thromboembolism
Keywords: unstable angina; acute coronary syndrome; fondaparinux sodium; non ST segment elevation myocardial infarction; myocardial infarction
MeSH Terms: conditions — Thromboembolism; Angina, Unstable; Acute Coronary Syndrome; Myocardial Infarction | interventions — Fondaparinux; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enoxaparin (Active Comparator)
  Interventions: Drug: enoxaparin
- Fondaparinux (Experimental)
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux — fondaparinux 2.5 mg, s.c. injection once daily x 8 days or Hospital Discharge if earlier and placebo-enoxaparin 1mg/kg s.c. injection twice daily x 2-8 days or until clinically stable
  Arms: Fondaparinux
Drug: enoxaparin — enoxaparin 1mg/kg s.c. injection twice daily x 2 to 8 days
  Arms: Enoxaparin

SUMMARY:
Study Objectives

PRIMARY OBJECTIVE: To evaluate whether fondaparinux is at least as effective as or superior to enoxaparin in preventing death, myocardial infarction or refactory ischemia up to Day 9 in the acute treatment of patients with unstable angina/non ST-segment elevation myocardial infarction concurrently managed with standard medical therapy.

SECONDARY OBJECTIVE: If non inferiority of fondaparinux is established on initial statistical analysis in a second step, superiority of fondaparinux to enoxaparin will be evaluated statistically.

* To determine whether fondaparinux is superior to enoxaparin in reducing death or MI at Day 9
* To determine whether fondaparinux is superior to enoxaparin in reducing major bleeding events up to Day 9
* To determine whether the relative effect on the primary end point of fondaparinux versus enoxaparin is sustained at Day 14, Day 30, Day 90 and Day 180

Study Drug: Patients will be randomized to receive either:

* Fondaparinux 2.5 mg once and placebo-enoxaparin twice daily by subcutaneous injection or
* Enoxaparin (1mg/kg) twice and fondaparinux-placebo once daily by subcutaneous injection

Duration of Therapy:

* Fondaparinux 2.5mg daily for 8 days or hospital discharge (whichever is earlier)
* Enoxaparin 1mg/kg b.i.d. x 2-8 days or until clinically stable.
* Patients should receive an ASA and all other standard medical therapies.

Substudy:

* A substudy comparing routine early coronary angiography immediately or as soon as possible (but no later than 24 hours after randomization) and intervention versus delayed (>48 hrs) coronary angiography and intervention.

Primary Outcome: The first occurence of any component of the following composite up to Day 9:

* Death
* Myocardial Infarction
* Refractory Ischemia

DETAILED DESCRIPTION:
This is a double-blind, double-dummy, randomized, parallel-group, controlled trial to compare the safety and efficacy of fondaparinux and enoxaparin in subjects with UA/NSTEMI (unstable angina/non ST segment myocardial infarction). Study drug (s.c.) was started immediately following randomization; subjects received fondaparinux 2.5mg once daily s.c for 8 days or until hospital discharge, if earlier, or enoxaparin 1mg/kg twice daily s.c for 2 to 8 days or until clinically stable. In subjects with creatinine clearance between 20mL/min and 30mL/min, enoxaparin was administered as 1mg/kg once daily. In addition to study drug, subjects were to receive standard medical care, including interventions (PCI [percutaneous coronary intervention] or coronary artery bypass graft surgery [CABG]).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting or admitted to hospital with symptoms suspected to represent an acute coronary syndrome.
* Able to randomize within 24 hours of the onset of the most recent episode of symptoms.
* At least one of the following additional criteria: (1) Troponin T of I or CK-MB above the upper limit of normal for the local institution and/or (2) ECG changes compatible with ischemia
* Written informed consent

Exclusion Criteria:

* Age < 21 years
* Any contraindication to low molecular weight heparin
* Hemorrhagic stroke within the last 12 months
* Indication for anticoagulation other than ACS.
* Pregnancy or women of childbearing potential who are not using an effective method of contraception
* Co-morbid condition with life expectancy less than 6 months
* Prior enrollment in one of the fondaparinux ACS trails or currently receiving an experimental pharmacologic agent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20078 (Actual)
Dates: Start 2003-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
death, myocardial infarction or refractory | up to and including Day 9
  first occurrence of any component of death, myocardial infarction or
major bleeding | Up to Day 9
  incidence of adjudicated major bleeding

SECONDARY OUTCOMES:
Death, myocardial infarction or refractory | up to Day 9, Day 14, Day 30,
  Incidence of the individual components of death, myocardial
major bleeding | up to and including Day 14, Day
  incidence of adjudicated major bleeding
Any bleeding (major or minor) | up to and including Day 9, Day
  Any bleeding (major or minor) as reported by the investigator as
Severe bleeding complications | up to and including Day 9, Day
  Severe bleeding complications according to modified thrombolysis in
Death, myocardial infarction | up to Days 9, 14, 30, 90 and
  composite of death, myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Fifth Organization to Assess Strategies in Acute Ischemic Syndromes Investigators; Yusuf S, Mehta SR, Chrolavicius S, Afzal R, Pogue J, Granger CB, Budaj A, Peters RJ, Bassand JP, Wallentin L, Joyner C, Fox KA. Comparison of fondaparinux and enoxaparin in acute coronary syndromes. N Engl J Med. 2006 Apr 6;354(14):1464-76. doi: 10.1056/NEJMoa055443. Epub 2006 Mar 14. PMID 16537663
- [Derived] Chow CK, Jolly S, Rao-Melacini P, Fox KA, Anand SS, Yusuf S. Association of diet, exercise, and smoking modification with risk of early cardiovascular events after acute coronary syndromes. Circulation. 2010 Feb 16;121(6):750-8. doi: 10.1161/CIRCULATIONAHA.109.891523. Epub 2010 Feb 1. PMID 20124123
- [Derived] Bassand JP, Afzal R, Eikelboom J, Wallentin L, Peters R, Budaj A, Fox KA, Joyner CD, Chrolavicius S, Granger CB, Mehta S, Yusuf S; OASIS 5 and OASIS 6 Investigators. Relationship between baseline haemoglobin and major bleeding complications in acute coronary syndromes. Eur Heart J. 2010 Jan;31(1):50-8. doi: 10.1093/eurheartj/ehp401. Epub 2009 Oct 12. PMID 19825809
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 103420 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103420 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 103420 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103420 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103420 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103420 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103420 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register